CLINICAL TRIAL: NCT03521765
Title: Occupational Therapy Interventions Based on Cancer Education on Quality of Life for Colorectal Cancer Survivors
Brief Title: Quality of Life in Colorectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Yang Shang-Yu, Mr., National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OTCRCQOL
Record Dates: First submitted 2018-04-29; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer
Keywords: quality of life; occupational therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT intervention group (Experimental): The OT intervention group were given a consultation based on a CRC education handbook by an occupational therapist for discharge preparation and on 1-month, 3-month follow-up clinic.
  Interventions: Other: Cancer education
- non-intervention group (No Intervention): The non-intervention group participants were given a CRC education handbook (the same handbook) only for discharge preparation.

INTERVENTIONS:
Other: Cancer education — Those participants in the OT intervention group were given a consultation based on a CRC education handbook by an occupational therapist for discharge preparation (about 30 minutes) and after each follow-up visit to the clinic (about 15-20 minutes); the non-intervention group participants were given a CRC education handbook (the same handbook) only for discharge preparation. For the first OT consultation, in the first 15 minutes, the occupational therapist educated the participants based on the CRC education handbook chapter by chapter. The next 15 minutes, the occupational therapist interacted with the participants and provided them customized lifestyle suggestions. For the each following (second and third) consultations, occupational therapists interacted with the participants and provided customized suggestions based on the participants' lifestyle at home.
  Arms: OT intervention group

SUMMARY:
BACKGROUND:

Colorectal cancer (CRC) and its treatment affect CRC survivors' quality of life (QoL), emotional distress and activities of daily living (ADL). It is assumed that occupational therapy interventions based on cancer education may be a feasible approach.

Aim To examine the effect of using cancer education based on healthy lifestyle by occupational therapist on QoL, emotional distress, ADL and healthy lifestyle behaviors in CRC survivors.

Methods Participants with CRC were designed as a two-group controlled trial, and a single-blind randomized controlled trial was conducted. These participants were randomly assigned to either an OT intervention or a non-intervention group (in a 1:1 ratio). Those participants in the OT intervention group were given a consultation based on a CRC education handbook by an occupational therapist for discharge preparation and on 1-month, 3-month follow-up clinic; the non-intervention group participants were given a CRC education handbook (the same handbook) only for discharge preparation. The primary outcome was the change in QoL measured using WHOOQOL-BREF. Secondary outcomes were changes in emotional distress, ADL and healthy lifestyle behaviors. Outcomes were examined in baseline (discharge preparation), 1-month and 3-months follow-up clinic.

ELIGIBILITY:
Inclusion Criteria:

* (1) had a new diagnosis of CRC and were suffering from cancer for the first time, (2) had undergone CRC hospitalization (surgical) treatments, (3) were able to communicate in Mandarin or Taiwanese.

Exclusion Criteria:

* Participants re-admitted within three months after discharge were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF(the World Health Organization Quality of Life-BREF) | 10 min
  The WHOQOL-BREF questionnaire is a self-assessment instrument, which is has been translated into several languages (The WHOQOL Group, 1998). It includes four domains: physical health, psychological health, social relationships, and environment.

SECONDARY OUTCOMES:
Brief Symptom Rating Scale (BSRS-5) | 3 min
  The Brief Symptom Rating Scale (BSRS-5) is used for screening psychiatric symptoms, which is to be able to quickly understand the psychological care needs of subjects. This scale includes only five items (anxiety, hostility, depression, low self-esteem, and insomnia), thus, the administration time is short.
Barthel Index (BI) | 5 min
  The Barthel Index (BI) measure the patients' performance on 10 ADL functions, and is commonly used scales which assess disability or dependence in activities of daily living for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, No.138,Sheng Li Road, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang SY, Wang JD, Chang JH. Occupational therapy to improve quality of life for colorectal cancer survivors: a randomized clinical trial. Support Care Cancer. 2020 Mar;28(3):1503-1511. doi: 10.1007/s00520-019-04971-2. Epub 2019 Jul 4. PMID 31273505